CLINICAL TRIAL: NCT02577341
Title: A Prospective Randomized Phase Ⅱ Study of Nimotuzumab Combined With Chemoradiotherapy for Unresectable, Locally Advanced Squamous Cell Lung Cancer
Brief Title: Nimotuzumab Combined With Chemoradiotherapy for Unresectable Locally Advanced Squamous Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-FXY-061
Record Dates: First submitted 2015-10-12; First posted 2015-10-16 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Non-small-cell Lung Cancer
Keywords: Nimotuzumab, Chemoradiotherapy,Squamous Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — nimotuzumab; Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nimotuzumab (Experimental): Daily RT to the chest, concurrent chemotherapy of weekly docetaxel and cisplatin, and concurrent weekly Nimotuzumab.
  Interventions: Drug: Nimotuzumab; Drug: docetaxel and cisplatin; Radiation: daily RT to the chest
- Control (Active Comparator): Daily RT to the chest, concurrent chemotherapy of weekly docetaxel and cisplatin.
  Interventions: Drug: docetaxel and cisplatin; Radiation: daily RT to the chest

INTERVENTIONS:
Drug: Nimotuzumab — Patients received weekly nimotuzumab (200mg, IV) concurrent with chemoradiotherapy.
  Arms: Nimotuzumab
Drug: docetaxel and cisplatin — Patients received weekly docetaxel and cisplatin, each of 1 day's duration,concurrent with chest radiotherapy
Radiation: daily RT to the chest — Patients received daily RT to the chest

SUMMARY:
This Phase II randomized study is to determine the efficacy and toxicity of Nimotuzumab in combined with chemoradiotherapy for unresectable,local advanced squamous cell lung cancer.

DETAILED DESCRIPTION:
This Phase II randomized study is to determine the efficacy and toxicity of Nimotuzumab combined with chemoradiotherapy for unresectable,locally advanced squamous cell lung cancer.

All patients were planned to receive radical dose of chest radiation and concurrent chemotherapy of weekly docetaxel and cisplatin, each of 1 day's duration.

Nimotuzumab group was treated with weekly nimotuzumab (200mg, IV) combined with chemoradiotherapy, while control group was treated with chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed squamous cell lung cancer
* patients have measurable or evaluable lesions based on the Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* unresectable phase IIIA(N2) and IIIB lung cancer confirmed by CT or MRI
* ECOG performance status 0-1
* Previously treated with chemotherapy or treatment-naive
* no previous chest radiotherapy, immunotherapy or biotherapy.
* hemoglobin≥10 mg/dL, platelet≥100000/μL,absolute neutrophil count ≥1500/μL
* serum creatinine ≤1.25 times the upper normal limit(UNL), or creatinine clearance≥60 ml/min
* bilirubin ≤1.5 times UNL, AST（SGOT）≤2.5 times UNL ,ALT（SGPT）≤2.5 times UNL,alkaline phosphatase ≤5 times UNL
* FEV1 >0.8 L
* CB6 within normal limits
* patients and their family signed the informed consents

Exclusion Criteria:

* adenosquamous carcinoma
* previous or recent another malignancy, except for nonmelanoma skin cancer or cervical cancer in situ
* contraindication for chemotherapy
* women in pregnancy, lactation period, or no pregnancy test 14 days before the first dose
* women who has the probability of pregnancy without contraception
* tendency of hemorrhage
* in other clinical trials within 30 days
* addicted in drugs or alcohol, AIDS patients
* uncontrollable seizure or psychotic patients without self-control ability
* severe allergy or idiosyncrasy
* not suitable for this study judged by researchers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2015-08; Primary Completion 2020-06 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
overall survival | 3 years

SECONDARY OUTCOMES:
Objective Response Rate | 3 years
progression-free survival | 3 years
rate of grade 3-4 radiation esophagitis | 1 years
  rate of grade 3-4 radiation esophagitis as assessed by CTCAE v4.0
rate of grade 3-4 radiation pneumonitis | 1 year
  rate of grade 3-4 radiation pneumonitis as assessed by CTCAE v4.0
Failure patterns | 3 years
  rates of local-regional recurrence, distant metastasis and brain metastasis

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Professor, Principal Investigator — Sun yat-sen universtiy cancer center
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Steel GG, Hill RP, Peckham MJ. Combined radiotherapy--chemotherapy of Lewis lung carcinoma. Int J Radiat Oncol Biol Phys. 1978 Jan-Feb;4(1-2):49-52. doi: 10.1016/0360-3016(78)90114-1. No abstract available. PMID 632147
- [Background] Chemotherapy in non-small cell lung cancer: a meta-analysis using updated data on individual patients from 52 randomised clinical trials. Non-small Cell Lung Cancer Collaborative Group. BMJ. 1995 Oct 7;311(7010):899-909. PMID 7580546
- [Background] Marino P, Preatoni A, Cantoni A. Randomized trials of radiotherapy alone versus combined chemotherapy and radiotherapy in stages IIIa and IIIb nonsmall cell lung cancer. A meta-analysis. Cancer. 1995 Aug 15;76(4):593-601. doi: 10.1002/1097-0142(19950815)76:43.0.co;2-n. PMID 8625152
- [Background] Pritchard RS, Anthony SP. Chemotherapy plus radiotherapy compared with radiotherapy alone in the treatment of locally advanced, unresectable, non-small-cell lung cancer. A meta-analysis. Ann Intern Med. 1996 Nov 1;125(9):723-9. doi: 10.7326/0003-4819-125-9-199611010-00003. PMID 8929005
- [Background] Kubota K, Furuse K, Kawahara M, Kodama N, Yamamoto M, Ogawara M, Negoro S, Masuda N, Takada M, Matsui K, et al. Role of radiotherapy in combined modality treatment of locally advanced non-small-cell lung cancer. J Clin Oncol. 1994 Aug;12(8):1547-52. doi: 10.1200/JCO.1994.12.8.1547. PMID 8040666
- [Background] Clinical practice guidelines for the treatment of unresectable non-small-cell lung cancer. Adopted on May 16, 1997 by the American Society of Clinical Oncology. J Clin Oncol. 1997 Aug;15(8):2996-3018. doi: 10.1200/JCO.1997.15.8.2996. PMID 9256144
- [Background] Stanley KE. Prognostic factors for survival in patients with inoperable lung cancer. J Natl Cancer Inst. 1980 Jul;65(1):25-32. PMID 6930515
- [Background] Mornex F, Houtte PV, Scalliet P, Loubeyre P. [Radiotherapy for non-small-cell bronchial cancers: definitions of volumes, patient selection. Recommendations of the International Association for the Study of Lung Cancer (IASLC)]. Cancer Radiother. 1998 Sep-Oct;2(5):579-89. doi: 10.1016/s1278-3218(98)80091-7. French. PMID 9868404
- [Background] Paesmans M, Sculier JP, Libert P, Bureau G, Dabouis G, Thiriaux J, Michel J, Van Cutsem O, Sergysels R, Mommen P, et al. Prognostic factors for survival in advanced non-small-cell lung cancer: univariate and multivariate analyses including recursive partitioning and amalgamation algorithms in 1,052 patients. The European Lung Cancer Working Party. J Clin Oncol. 1995 May;13(5):1221-30. doi: 10.1200/JCO.1995.13.5.1221. PMID 7738625
- [Background] Scott C, Sause WT, Byhardt R, Marcial V, Pajak TF, Herskovic A, Cox JD. Recursive partitioning analysis of 1592 patients on four Radiation Therapy Oncology Group studies in inoperable non-small cell lung cancer. Lung Cancer. 1997 Jun;17 Suppl 1:S59-74. doi: 10.1016/s0169-5002(97)00640-5. PMID 9213303
- [Background] Curran WJ, Scott C, Langer C, et al. Phase III comoarision of sequential vs concurrent chemoradiation therapy for patients with unresectable stage III non-small cell lung cancer: initial report of RTOG 9410. Proc Am Soc Clin Oncol, 2000, 19: 484a.
- [Background] Furuse K, Fukuoka M, Kawahara M, Nishikawa H, Takada Y, Kudoh S, Katagami N, Ariyoshi Y. Phase III study of concurrent versus sequential thoracic radiotherapy in combination with mitomycin, vindesine, and cisplatin in unresectable stage III non-small-cell lung cancer. J Clin Oncol. 1999 Sep;17(9):2692-9. doi: 10.1200/JCO.1999.17.9.2692. PMID 10561343
- [Background] Auperin A, Le Pechoux C, Rolland E, Curran WJ, Furuse K, Fournel P, Belderbos J, Clamon G, Ulutin HC, Paulus R, Yamanaka T, Bozonnat MC, Uitterhoeve A, Wang X, Stewart L, Arriagada R, Burdett S, Pignon JP. Meta-analysis of concomitant versus sequential radiochemotherapy in locally advanced non-small-cell lung cancer. J Clin Oncol. 2010 May 1;28(13):2181-90. doi: 10.1200/JCO.2009.26.2543. Epub 2010 Mar 29. PMID 20351327
- [Background] Pfister DG, Johnson DH, Azzoli CG, Sause W, Smith TJ, Baker S Jr, Olak J, Stover D, Strawn JR, Turrisi AT, Somerfield MR; American Society of Clinical Oncology. American Society of Clinical Oncology treatment of unresectable non-small-cell lung cancer guideline: update 2003. J Clin Oncol. 2004 Jan 15;22(2):330-53. doi: 10.1200/JCO.2004.09.053. Epub 2003 Dec 22. No abstract available. PMID 14691125
- [Background] Ardizzoni A, Tiseo M, Boni L et al. CISCA (cis-platin vs. carboplatin) meta-analysis: an individual patient data meta-analysis comparing cisplatin versus carboplatin-based chemotherapy in first-line treatment of advanced non-small cell lung cancer (NSCLC) [Abstract 7011]. Proc AmSoc Clin Oncol 2006;24:366S.
- [Background] Rosell R, Moran T, Queralt C, Porta R, Cardenal F, Camps C, Majem M, Lopez-Vivanco G, Isla D, Provencio M, Insa A, Massuti B, Gonzalez-Larriba JL, Paz-Ares L, Bover I, Garcia-Campelo R, Moreno MA, Catot S, Rolfo C, Reguart N, Palmero R, Sanchez JM, Bastus R, Mayo C, Bertran-Alamillo J, Molina MA, Sanchez JJ, Taron M; Spanish Lung Cancer Group. Screening for epidermal growth factor receptor mutations in lung cancer. N Engl J Med. 2009 Sep 3;361(10):958-67. doi: 10.1056/NEJMoa0904554. Epub 2009 Aug 19. PMID 19692684
- [Background] Mok TS, Wu YL, Thongprasert S, Yang CH, Chu DT, Saijo N, Sunpaweravong P, Han B, Margono B, Ichinose Y, Nishiwaki Y, Ohe Y, Yang JJ, Chewaskulyong B, Jiang H, Duffield EL, Watkins CL, Armour AA, Fukuoka M. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. PMID 19692680
- [Background] Maemondo M, Inoue A, Kobayashi K, Sugawara S, Oizumi S, Isobe H, Gemma A, Harada M, Yoshizawa H, Kinoshita I, Fujita Y, Okinaga S, Hirano H, Yoshimori K, Harada T, Ogura T, Ando M, Miyazawa H, Tanaka T, Saijo Y, Hagiwara K, Morita S, Nukiwa T; North-East Japan Study Group. Gefitinib or chemotherapy for non-small-cell lung cancer with mutated EGFR. N Engl J Med. 2010 Jun 24;362(25):2380-8. doi: 10.1056/NEJMoa0909530. PMID 20573926
- [Background] Kwak EL, Bang YJ, Camidge DR, Shaw AT, Solomon B, Maki RG, Ou SH, Dezube BJ, Janne PA, Costa DB, Varella-Garcia M, Kim WH, Lynch TJ, Fidias P, Stubbs H, Engelman JA, Sequist LV, Tan W, Gandhi L, Mino-Kenudson M, Wei GC, Shreeve SM, Ratain MJ, Settleman J, Christensen JG, Haber DA, Wilner K, Salgia R, Shapiro GI, Clark JW, Iafrate AJ. Anaplastic lymphoma kinase inhibition in non-small-cell lung cancer. N Engl J Med. 2010 Oct 28;363(18):1693-703. doi: 10.1056/NEJMoa1006448. PMID 20979469
- [Background] Schiller JH, Harrington D, Belani CP, Langer C, Sandler A, Krook J, Zhu J, Johnson DH; Eastern Cooperative Oncology Group. Comparison of four chemotherapy regimens for advanced non-small-cell lung cancer. N Engl J Med. 2002 Jan 10;346(2):92-8. doi: 10.1056/NEJMoa011954. PMID 11784875
- [Background] Sandler A, Gray R, Perry MC, Brahmer J, Schiller JH, Dowlati A, Lilenbaum R, Johnson DH. Paclitaxel-carboplatin alone or with bevacizumab for non-small-cell lung cancer. N Engl J Med. 2006 Dec 14;355(24):2542-50. doi: 10.1056/NEJMoa061884. PMID 17167137
- [Background] Pao W, Miller V, Zakowski M, Doherty J, Politi K, Sarkaria I, Singh B, Heelan R, Rusch V, Fulton L, Mardis E, Kupfer D, Wilson R, Kris M, Varmus H. EGF receptor gene mutations are common in lung cancers from "never smokers" and are associated with sensitivity of tumors to gefitinib and erlotinib. Proc Natl Acad Sci U S A. 2004 Sep 7;101(36):13306-11. doi: 10.1073/pnas.0405220101. Epub 2004 Aug 25. PMID 15329413
- [Background] Paez JG, Janne PA, Lee JC, Tracy S, Greulich H, Gabriel S, Herman P, Kaye FJ, Lindeman N, Boggon TJ, Naoki K, Sasaki H, Fujii Y, Eck MJ, Sellers WR, Johnson BE, Meyerson M. EGFR mutations in lung cancer: correlation with clinical response to gefitinib therapy. Science. 2004 Jun 4;304(5676):1497-500. doi: 10.1126/science.1099314. Epub 2004 Apr 29. PMID 15118125
- [Background] Lynch TJ, Bell DW, Sordella R, Gurubhagavatula S, Okimoto RA, Brannigan BW, Harris PL, Haserlat SM, Supko JG, Haluska FG, Louis DN, Christiani DC, Settleman J, Haber DA. Activating mutations in the epidermal growth factor receptor underlying responsiveness of non-small-cell lung cancer to gefitinib. N Engl J Med. 2004 May 20;350(21):2129-39. doi: 10.1056/NEJMoa040938. Epub 2004 Apr 29. PMID 15118073
- [Background] Sun Y, Ren Y, Fang Z, Li C, Fang R, Gao B, Han X, Tian W, Pao W, Chen H, Ji H. Lung adenocarcinoma from East Asian never-smokers is a disease largely defined by targetable oncogenic mutant kinases. J Clin Oncol. 2010 Oct 20;28(30):4616-20. doi: 10.1200/JCO.2010.29.6038. Epub 2010 Sep 20. PMID 20855837
- [Background] Pirker R, Pereira JR, Szczesna A, von Pawel J, Krzakowski M, Ramlau R, Vynnychenko I, Park K, Yu CT, Ganul V, Roh JK, Bajetta E, O'Byrne K, de Marinis F, Eberhardt W, Goddemeier T, Emig M, Gatzemeier U; FLEX Study Team. Cetuximab plus chemotherapy in patients with advanced non-small-cell lung cancer (FLEX): an open-label randomised phase III trial. Lancet. 2009 May 2;373(9674):1525-31. doi: 10.1016/S0140-6736(09)60569-9. PMID 19410716
- [Background] Weiss J, Sos ML, Seidel D, Peifer M, Zander T, Heuckmann JM, Ullrich RT, Menon R, Maier S, Soltermann A, Moch H, Wagener P, Fischer F, Heynck S, Koker M, Schottle J, Leenders F, Gabler F, Dabow I, Querings S, Heukamp LC, Balke-Want H, Ansen S, Rauh D, Baessmann I, Altmuller J, Wainer Z, Conron M, Wright G, Russell P, Solomon B, Brambilla E, Brambilla C, Lorimier P, Sollberg S, Brustugun OT, Engel-Riedel W, Ludwig C, Petersen I, Sanger J, Clement J, Groen H, Timens W, Sietsma H, Thunnissen E, Smit E, Heideman D, Cappuzzo F, Ligorio C, Damiani S, Hallek M, Beroukhim R, Pao W, Klebl B, Baumann M, Buettner R, Ernestus K, Stoelben E, Wolf J, Nurnberg P, Perner S, Thomas RK. Frequent and focal FGFR1 amplification associates with therapeutically tractable FGFR1 dependency in squamous cell lung cancer. Sci Transl Med. 2010 Dec 15;2(62):62ra93. doi: 10.1126/scitranslmed.3001451. PMID 21160078
- [Background] Sos ML, Michel K, Zander T, Weiss J, Frommolt P, Peifer M, Li D, Ullrich R, Koker M, Fischer F, Shimamura T, Rauh D, Mermel C, Fischer S, Stuckrath I, Heynck S, Beroukhim R, Lin W, Winckler W, Shah K, LaFramboise T, Moriarty WF, Hanna M, Tolosi L, Rahnenfuhrer J, Verhaak R, Chiang D, Getz G, Hellmich M, Wolf J, Girard L, Peyton M, Weir BA, Chen TH, Greulich H, Barretina J, Shapiro GI, Garraway LA, Gazdar AF, Minna JD, Meyerson M, Wong KK, Thomas RK. Predicting drug susceptibility of non-small cell lung cancers based on genetic lesions. J Clin Invest. 2009 Jun;119(6):1727-40. doi: 10.1172/JCI37127. Epub 2009 May 18. PMID 19451690
- [Background] Sos ML, Fischer S, Ullrich R, Peifer M, Heuckmann JM, Koker M, Heynck S, Stuckrath I, Weiss J, Fischer F, Michel K, Goel A, Regales L, Politi KA, Perera S, Getlik M, Heukamp LC, Ansen S, Zander T, Beroukhim R, Kashkar H, Shokat KM, Sellers WR, Rauh D, Orr C, Hoeflich KP, Friedman L, Wong KK, Pao W, Thomas RK. Identifying genotype-dependent efficacy of single and combined PI3K- and MAPK-pathway inhibition in cancer. Proc Natl Acad Sci U S A. 2009 Oct 27;106(43):18351-6. doi: 10.1073/pnas.0907325106. Epub 2009 Oct 5. PMID 19805051
- [Background] Marek L, Ware KE, Fritzsche A, Hercule P, Helton WR, Smith JE, McDermott LA, Coldren CD, Nemenoff RA, Merrick DT, Helfrich BA, Bunn PA Jr, Heasley LE. Fibroblast growth factor (FGF) and FGF receptor-mediated autocrine signaling in non-small-cell lung cancer cells. Mol Pharmacol. 2009 Jan;75(1):196-207. doi: 10.1124/mol.108.049544. Epub 2008 Oct 10. PMID 18849352
- [Background] Mendelsohn J. Targeting the epidermal growth factor receptor for cancer therapy. J Clin Oncol. 2002 Sep 15;20(18 Suppl):1S-13S. No abstract available. PMID 12235219
- [Background] Mendelsohn J. Epidermal growth factor receptor inhibition by a monoclonal antibody as anticancer therapy. Clin Cancer Res. 1997 Dec;3(12 Pt 2):2703-7. PMID 10068277
- [Background] Deonarain MP, Kousparou CA, Epenetos AA. Antibodies targeting cancer stem cells: a new paradigm in immunotherapy? MAbs. 2009 Jan-Feb;1(1):12-25. doi: 10.4161/mabs.1.1.7347. PMID 20046569
- [Background] Dragovich T, Campen C. Anti-EGFR-Targeted Therapy for Esophageal and Gastric Cancers: An Evolving Concept. J Oncol. 2009;2009:804108. doi: 10.1155/2009/804108. Epub 2009 Jul 14. PMID 19636422
- [Background] Essack M, Radovanovic A, Schaefer U, Schmeier S, Seshadri SV, Christoffels A, Kaur M, Bajic VB. DDEC: Dragon database of genes implicated in esophageal cancer. BMC Cancer. 2009 Jul 6;9:219. doi: 10.1186/1471-2407-9-219. PMID 19580656
- [Background] Jimeno A, Messersmith WA, Hirsch FR, Franklin WA, Eckhardt SG. KRAS mutations and sensitivity to epidermal growth factor receptor inhibitors in colorectal cancer: practical application of patient selection. J Clin Oncol. 2009 Mar 1;27(7):1130-6. doi: 10.1200/JCO.2008.19.8168. Epub 2009 Jan 5. PMID 19124802
- [Background] Mukohara T, Engelman JA, Hanna NH, Yeap BY, Kobayashi S, Lindeman N, Halmos B, Pearlberg J, Tsuchihashi Z, Cantley LC, Tenen DG, Johnson BE, Janne PA. Differential effects of gefitinib and cetuximab on non-small-cell lung cancers bearing epidermal growth factor receptor mutations. J Natl Cancer Inst. 2005 Aug 17;97(16):1185-94. doi: 10.1093/jnci/dji238. PMID 16106023
- [Background] Akashi Y, Okamoto I, Iwasa T, Yoshida T, Suzuki M, Hatashita E, Yamada Y, Satoh T, Fukuoka M, Ono K, Nakagawa K. Enhancement of the antitumor activity of ionising radiation by nimotuzumab, a humanised monoclonal antibody to the epidermal growth factor receptor, in non-small cell lung cancer cell lines of differing epidermal growth factor receptor status. Br J Cancer. 2008 Feb 26;98(4):749-55. doi: 10.1038/sj.bjc.6604222. Epub 2008 Feb 5. PMID 18253126
- [Background] 林凤武等, 相近分化的肺鳞癌和腺癌中PCNA及EGFR表达的研究. 白求恩医科大学学报, 2000. 26(4): 第358-360页
- [Background] Eropean organization for research and treatment of cancer. EORTC QLQ-OES18. Available from: http://groups.eortc.be/qol/downloads/modules/specimen_20qlq_oes18.pdf 42.
- [Background] Solit DB, Rosen N. Hsp90: a novel target for cancer therapy. Curr Top Med Chem. 2006;6(11):1205-14. doi: 10.2174/156802606777812068. PMID 16842157
- [Background] Giezen TJ, Mantel-Teeuwisse AK, Straus SM, Schellekens H, Leufkens HG, Egberts AC. Safety-related regulatory actions for biologicals approved in the United States and the European Union. JAMA. 2008 Oct 22;300(16):1887-96. doi: 10.1001/jama.300.16.1887. PMID 18940975
- [Background] 2012 ASCO Annual Meeting, J Clin Oncol 30, 2012 (suppl; abstr e14604)
- [Background] Bebb G, Smith C, Rorke S, Boland W, Nicacio L, Sukhoo R, Brade A. Phase I clinical trial of the anti-EGFR monoclonal antibody nimotuzumab with concurrent external thoracic radiotherapy in Canadian patients diagnosed with stage IIb, III or IV non-small cell lung cancer unsuitable for radical therapy. Cancer Chemother Pharmacol. 2011 Apr;67(4):837-45. doi: 10.1007/s00280-010-1379-9. Epub 2010 Jun 20. PMID 20563810
- [Background] Choi HJ, Sohn JH, Lee CG, Shim HS, Lee IJ, Yang WI, Kwon JE, Kim SK, Park MS, Lee JH, Kim JH. A phase I study of nimotuzumab in combination with radiotherapy in stages IIB-IV non-small cell lung cancer unsuitable for radical therapy: Korean results. Lung Cancer. 2011 Jan;71(1):55-9. doi: 10.1016/j.lungcan.2010.04.010. Epub 2010 May 7. PMID 20451284
- [Background] Li LF, Wang HQ, Liu XM, Zhang HL, Qiu LH, Qian ZZ, Li W. [Nimotuzumab in combination with chemotherapy in patients with advanced non-small cell lung cancer]. Zhonghua Zhong Liu Za Zhi. 2011 Aug;33(8):626-8. Chinese. PMID 22325226
- [Background] Babu KG, Prabhash K, Vaid AK, Sirohi B, Diwakar RB, Rao R, Kar M, Malhotra H, Nag S, Goswami C, Raina V, Mohan R. Nimotuzumab plus chemotherapy versus chemotherapy alone in advanced non-small-cell lung cancer: a multicenter, randomized, open-label Phase II study. Onco Targets Ther. 2014 Jun 13;7:1051-60. doi: 10.2147/OTT.S63168. eCollection 2014. PMID 24966687